CLINICAL TRIAL: NCT00972478
Title: A Phase I/II Trial of Vorinostat (SAHA) (NSC-701852) in Combination With Rituximab-CHOP in Patients With Newly Diagnosed Advanced Stage Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Vorinostat, Rituximab, and Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage II, Stage III, or Stage IV Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01964; NCI-2011-01964 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000653803; S0806 (Other: SWOG); S0806 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Ann Arbor Stage II Non-Hodgkin Lymphoma; Ann Arbor Stage III Non-Hodgkin Lymphoma; Ann Arbor Stage IV Non-Hodgkin Lymphoma
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive vorinostat PO once daily on days 1-5 or 1-9 (according to dose level), rituximab IV, cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 3. Patients also receive prednisone PO once daily on days 3-7. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate; Drug: Vorinostat

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given IV
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I/II trial is studying the side effects and best dose of vorinostat when given together with rituximab and combination chemotherapy and to see how well it works in treating patients with newly diagnosed stage II, stage III, or stage IV diffuse large B-cell lymphoma. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cell-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with rituximab and combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To find a safe dose of vorinostat to be used in combination with R-CHOP (rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone) (vorinostat-R-CHOP). (Phase I) II. To estimate the 2-year progression-free survival (PFS) rate in patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL) treated with vorinostat and R-CHOP therapy (vorinostat-R-CHOP). (Phase II) III. To estimate the response rate (complete and partial) and 2-year overall survival rate. (Phase II) IV. To evaluate the toxicity of vorinostat-R-CHOP in patients with newly diagnosed DLBCL. (Phase II) V. To assess whether pre-treatment acetylation status of histones, expression of major histocompatibility complex (MHC) class II genes, and/or percentage of cluster of differentiation (CD)8+ tumor infiltrating lymphocytes correlate with progression-free survival. (Phase II) VI. To explore whether treatment with vorinostat-R-CHOP increases histone acetylation, alters expression of MHC class II proteins, or alters percentage of T-cell subsets (CD8+, CD4+, forkhead box P3 [FOXP3]+) or infiltrating macrophages. (Phase II) VII. To explore whether histone acetylation status of tumor tissues correlates with MHC class II expression of peripheral blood B cells and lymphocyte subsets. (Phase II) VIII. To explore whether the change in systemic levels of immune cytokines with vorinostat-R-CHOP correlates with lymphoma symptoms, response, progression-free or overall survival. (Phase II)

OUTLINE: This is a phase I, dose escalation study of vorinostat followed by a phase II study.

Patients receive vorinostat orally (PO) once daily on days 1-5 or 1-9 (according to dose level), rituximab intravenously (IV), cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 3. Patients also receive prednisone PO once daily on days 3-7. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for 2 years, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy proven, newly diagnosed DLBCL with stage II bulky, stage III or stage IV disease, with an International Prognostic Index (IPI) or revised (R)-IPI score greater than 0; a report providing confirmation of CD20 expression must be submitted
* Adequate sections from the original diagnostic specimen must be available for submission for review by the Southwest Oncology Group (SWOG) Lymphoma Pathology Laboratory; an adequate biopsy requires sufficient tissue to establish the architecture and World Health Organization (WHO) histologic subtype with certainty; fine needle aspiration or cytology is not adequate
* Patients must be offered the opportunity to consent to the correlative science studies; patients are encouraged to submit specimens for correlative studies; however, specimen submission is not a requirement for participation in the study
* Patients must have measurable disease; measurable disease must be determined by computed tomography (CT) scan of chest, abdomen and pelvis performed within 28 days prior to registration; positron emission tomography (PET)/CT may be substituted for CT scan only if CT scan is of diagnostic quality and is contrast enhanced
* Patients must have a unilateral bone marrow aspirate and biopsy for staging performed within 42 days prior to registration
* Patients must not have clinical evidence of central nervous system involvement by lymphoma; any laboratory or radiographic tests performed within 42 days prior to registration to assess central nervous system (CNS) involvement must be negative
* Patients must not have received prior chemotherapy, radiation, or antibody therapy for lymphoma; steroid pre-medication for IV contrast allergy is allowed
* Patients must have Zubrod performance status of 0-2
* Patients must have serum lactate dehydrogenase (LDH) measured within 28 days prior to registration
* Absolute neutrophil count (ANC) > 1,000/mcL within 28 days prior to registration, unless due to bone marrow infiltration by lymphoma
* Platelets > 100,000/mcL within 28 days prior to registration, unless due to bone marrow infiltration by lymphoma
* Cardiac ejection fraction ≥ institutional lower limit of normal (ILLN) by multigated acquisition (MUGA) scan or 2-dimensional (2-D) echocardiogram (ECHO) with no significant abnormalities within 42 days prior to registration
* Patients must not have received valproic acid (a histone deacetylase [HDAC] inhibitor) within 28 days prior to registration
* Patients must have no known hypersensitivity to the components of treatment
* Patients must be willing to discontinue taking any medications that are generally accepted to have a risk of causing Torsades de Pointes while on study
* Patients known to be human immunodeficiency virus (HIV) positive are not eligible; existing therapeutic options are effective and study design does not support assessing the efficacy of treatment on those with HIV
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2026-03-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Persky, Principal Investigator — SWOG Cancer Research Network
Locations (190):
- United States (190):
  - Providence Hospital, Mobile, Alabama
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Yale University, New Haven, Connecticut
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - DeSoto Regional Health System, Mansfield, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Overton Brooks Veteran's Administration Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Saint Charles Health System, Bend, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Ph I: R-CHOP+Vorinostat (400mg D1-9): Patients receive vorinostat 400 mg PO once daily on days 1-9 (according to dose level), rituximab IV, cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 3. Patients also receive prednisone PO once daily on days 3-7. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
- Ph II: R-CHOP+Vorinostat: Patients receive vorinostat 400 mg PO once daily on days 1-5 or 1-9 (according to dose level), rituximab IV, cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 3. Patients also receive prednisone PO once daily on days 3-7. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ph I: R-CHOP+Vorinostat (400mg D1-9) | Ph II: R-CHOP+Vorinostat
Started | 11 | 72
Eligible and Began Protocol Therapy | 9 | 63
Completed | 4 | 34
Not Completed | 7 | 38
Not completed — Adverse Event | 3 | 16
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Progression/Relapse | 0 | 2
Not completed — Death | 0 | 2
Not completed — Not protocol specified | 1 | 1
Not completed — Ineligible | 1 | 7
Not completed — Not start protocol treatment | 1 | 2

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph I: R-CHOP+Vorinostat (400mg D1-9) | Ph II: R-CHOP+Vorinostat | Total
Number analyzed (Participants) | 9 | 63 | 72
Age, Continuous [Median (Full Range); unit: years] | 66.9 [46.4 to 83.8] | 64.1 [19.6 to 80.8] | 64.2 [19.6 to 83.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 27 | 30
  Male | 6 | 36 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9 | 54 | 63
  Black | 0 | 3 | 3
  Asian | 0 | 5 | 5
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 3 | 4 | 7
  Non-Hispanic | 6 | 59 | 65

OUTCOME MEASURES:

1. Primary Outcome: Safe Dose of Vorinostat to be Used in Combination With R-CHOP Assessed by CTCAE Version 4.0 (Phase I)
Description: Safe dose of Vorinostat (in combination with R-CHOP) at which 3/10 or fewer patients have doselimiting toxicities (DLT). Toxicities graded according to the NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0). DLT apply only during cycle 1 and should be drug-related (possible, probable, or definite).
Time Frame: 21 days
Population: Phase I eligible patients receiving any amount of the assigned dose during Cycle 1 (1 Cycle = 21 days) or whom developed a dose-limiting toxicity (DLT).
Measure: Number; unit: mg PO Once daily Days 1-9
Arm/Group | Ph I: R-CHOP+Vorinostat (400mg D1-9)
Number analyzed (Participants) | 9
mg PO Once daily Days 1-9 | 400

2. Primary Outcome: Progression-free Survival (Phase II)
Description: From date of registration to date of first documentation of progressive disease, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Up to 2 years
Population: Eligible patients who received the protocol treatment in the Phase II portion of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ph II: R-CHOP+Vorinostat
Number analyzed (Participants) | 63
percentage of participants | 73 [59.6 to 81.9]

3. Secondary Outcome: Overall Survival (Phase II)
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 2 years
Population: Eligible patients who received the protocol treatment in the Phase II portion of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ph II: R-CHOP+Vorinostat
Number analyzed (Participants) | 63
percentage of participants | 86 [74.3 to 92.3]

4. Secondary Outcome: Response Rate (Complete Response [CR]+Partial Response [PR]) (Phase II)
Description: Objective disease status is evaluated according to the 2007 revised Cheson et al. criteria. Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow (BM) must be negative if positive at baseline. Normalization of markers. Partial Response (PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: Up to week 26
Population: Eligible patients who received the protocol treatment in the Phase II portion of the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ph II: R-CHOP+Vorinostat
Number analyzed (Participants) | 63
percentage of participants | 81 [69.1 to 89.8]

5. Secondary Outcome: Toxicity of Vorinostat-R-CHOP in Patients With Newly Diagnosed DLBCL
Description: Incidence of toxicity as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Up to week 26
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Ph I: R-CHOP+Vorinostat (400mg D1-9) | Ph II: R-CHOP+Vorinostat
Number analyzed (Participants) | 9 | 63
Participants
  Abdominal pain | 1 | 3
  Acute kidney injury | 0 | 1
  Alanine aminotransferase increased | 0 | 1
  Anemia | 4 | 22
  Anorexia | 1 | 2
  Aspartate aminotransferase increased | 0 | 1
  Atrial fibrillation | 0 | 1
  Bladder spasm | 0 | 1
  Bronchial infection | 0 | 1
  CD4 lymphocytes decreased | 0 | 1
  CPK increased | 0 | 1
  Carbon monoxide diffusing capacity decreased | 0 | 1
  Colitis | 1 | 0
  Creatinine increased | 1 | 0
  Cystitis noninfective | 0 | 1
  Dehydration | 2 | 4
  Depression | 1 | 0
  Diarrhea | 2 | 2
  Disseminated intravascular coagulation | 1 | 0
  Dizziness | 1 | 0
  Duodenal perforation | 0 | 1
  Dysphagia | 0 | 1
  Dyspnea | 0 | 1
  Electrocardiogram QT corrected interval prolonged | 1 | 1
  Fatigue | 3 | 9
  Febrile neutropenia | 3 | 24
  Fecal incontinence | 0 | 1
  Gastrointestinal disorders - Other, specify | 0 | 1
  Generalized muscle weakness | 2 | 2
  Hematuria | 1 | 0
  Hiccups | 0 | 1
  Hyperglycemia | 0 | 4
  Hypoalbuminemia | 1 | 3
  Hypocalcemia | 1 | 0
  Hypokalemia | 2 | 8
  Hyponatremia | 0 | 6
  Hypophosphatemia | 1 | 2
  Hypotension | 0 | 3
  Infections and infestations - Other, specify | 1 | 3
  Jejunal perforation | 0 | 1
  Left ventricular systolic dysfunction | 0 | 1
  Leukocytosis | 0 | 1
  Lung infection | 0 | 4
  Lymphocyte count decreased | 4 | 20
  Mucosal infection | 0 | 1
  Mucositis oral | 1 | 3
  Multi-organ failure | 1 | 0
  Myalgia | 1 | 2
  Myocardial infarction | 0 | 2
  Nausea | 1 | 3
  Neutrophil count decreased | 8 | 37
  Obstruction gastric | 0 | 1
  Pain | 0 | 1
  Paronychia | 0 | 1
  Peripheral motor neuropathy | 1 | 0
  Platelet count decreased | 4 | 22
  Pneumonitis | 0 | 1
  Recurrent laryngeal nerve palsy | 0 | 1
  Respiratory failure | 0 | 1
  Sepsis | 3 | 11
  Sinus tachycardia | 0 | 1
  Sinusitis | 0 | 1
  Small intestinal obstruction | 0 | 1
  Stoma site infection | 0 | 1
  Syncope | 0 | 4
  Urinary tract infection | 0 | 3
  Urinary tract pain | 0 | 2
  Urine output decreased | 1 | 0
  Vasovagal reaction | 0 | 1
  Visceral arterial ischemia | 1 | 0
  Vomiting | 0 | 2
  Weight loss | 0 | 3
  White blood cell decreased | 7 | 32

ADVERSE EVENTS:
Time Frame: Up to week 26
Description: Eligible patients who had received any treatment were included. Incidence of toxicity as assessed by the Common Terminology Criteria for Adverse Events version 4.0.
Arm/Group | Ph I: R-CHOP+Vorinostat (400mg D1-9) | Ph II: R-CHOP+Vorinostat
Serious Adverse Events (participants affected / at risk) | 5/9 | 44/63
Other Adverse Events (participants affected / at risk) | 9/9 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ph I: R-CHOP+Vorinostat (400mg D1-9) (N=9) | Ph II: R-CHOP+Vorinostat (N=63)
Anemia (Blood and lymphatic system disorders) | 3 | 13
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 22
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 2
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 3
Fever (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 4
Paronychia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 8
Sinusitis (Infections and infestations) | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 4
Neutrophil count decreased (Investigations) | 3 | 16
Platelet count decreased (Investigations) | 4 | 16
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 2 | 10
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Confusion (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 3
Thromboembolic event (Vascular disorders) | 0 | 2
Visceral arterial ischemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ph I: R-CHOP+Vorinostat (400mg D1-9) (N=9) | Ph II: R-CHOP+Vorinostat (N=63)
Anemia (Blood and lymphatic system disorders) | 9 | 52
Sinus tachycardia (Cardiac disorders) | 0 | 9
Blurred vision (Eye disorders) | 2 | 8
Dry eye (Eye disorders) | 2 | 0
Eye disorders-Other (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Watering eyes (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 16
Bloating (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 5 | 26
Diarrhea (Gastrointestinal disorders) | 7 | 31
Dry mouth (Gastrointestinal disorders) | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Fecal incontinence (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 4
Mucositis oral (Gastrointestinal disorders) | 1 | 22
Nausea (Gastrointestinal disorders) | 8 | 43
Oral pain (Gastrointestinal disorders) | 1 | 2
Rectal mucositis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 22
Chills (General disorders) | 2 | 10
Edema face (General disorders) | 3 | 0
Edema limbs (General disorders) | 2 | 17
Fatigue (General disorders) | 8 | 45
Fever (General disorders) | 1 | 18
Gait disturbance (General disorders) | 2 | 3
Infusion related reaction (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 0 | 4
Pain (General disorders) | 4 | 7
Infections and infestations-Other (Infections and infestations) | 1 | 4
Mucosal infection (Infections and infestations) | 1 | 3
Peripheral nerve infection (Infections and infestations) | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 1 | 5
Wound infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 16
Alkaline phosphatase increased (Investigations) | 0 | 11
Aspartate aminotransferase increased (Investigations) | 2 | 13
Blood bilirubin increased (Investigations) | 1 | 4
CD4 lymphocytes decreased (Investigations) | 0 | 4
Cardiac troponin I increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 1 | 6
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 5
Investigations-Other (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 7 | 26
Neutrophil count decreased (Investigations) | 7 | 35
Platelet count decreased (Investigations) | 8 | 32
Urine output decreased (Investigations) | 1 | 0
Weight gain (Investigations) | 2 | 4
Weight loss (Investigations) | 2 | 13
White blood cell decreased (Investigations) | 8 | 40
Anorexia (Metabolism and nutrition disorders) | 6 | 23
Dehydration (Metabolism and nutrition disorders) | 2 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 20
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 20
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 4 | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 8
Hyponatremia (Metabolism and nutrition disorders) | 4 | 23
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 7
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 9
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 12
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 4 | 20
Dysgeusia (Nervous system disorders) | 3 | 8
Headache (Nervous system disorders) | 4 | 20
Lethargy (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Movements involuntary (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 5 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 19
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 9
Confusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 6 | 10
Hematuria (Renal and urinary disorders) | 1 | 4
Proteinuria (Renal and urinary disorders) | 0 | 7
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 6 | 5
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 21
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 5
Hypertension (Vascular disorders) | 4 | 11
Hypotension (Vascular disorders) | 2 | 8
Thromboembolic event (Vascular disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less